CLINICAL TRIAL: NCT05723653
Title: Harnessing Social Network Support to Improve Retention in Care and Viral Suppression Among People Living With HIV in Chicago and Alabama: A Hybrid Type I Effectiveness-implementation Trial
Brief Title: Hybrid Type I Effectiveness-Implementation Trial of a Social Network Support Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Tulane University (Other); University of Alabama at Birmingham (Other); Birmingham AIDS Outreach (Unknown); Chicago Center for HIV Elimination (Unknown); Howard Brown Health (Unknown); Thrive Alabama (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0110
Record Dates: First submitted 2023-01-30; First posted 2023-02-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-01

CONDITIONS: HIV Seropositivity
Keywords: HIV care engagement; HIV viral suppression; Social support; Social networks
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: Following study registration (at which a unique Study Identification (ID) will be assigned), Index participants will be randomized to either the intervention group (n=300) or Treatment as Usual (n=300). Intervention arm Indexes will identify a Support Confidant (SC) (creating Index-SC dyads). Study staff will discuss pros and cons of treatment as usual (equipoise induction) to balance the desirability of the two intervention conditions.
  After the 12-month follow-up survey, we will re-randomize the 300 Index-Support Confidant dyads in the intervention condition with equal probability to continue receiving standard mini-boosters (n=150 Index-Support Confidant dyads) or a return to treatment as usual (n=150 Index-Support Confidant dyads). The randomization schedule will be prepared in advance, and treatment assignment will be obtained using the randomization module in REDCap.
Masking Description: Due to the nature of the intervention, it is not possible to blind participants, interventionists, and investigators. However, we take the following steps to minimize bias, assess contamination, and enhance rigor: (1) collecting baseline data prior to randomization; (2) Treatment as Usual (TAU) providers are blinded to allocation; and (3) assessing contamination at follow-up surveys by identifying overlap between the networks of those in each study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Network Support Intervention Condition (Experimental): The intervention condition will be delivered by trained Intervention Case Managers to n=300 Index participants and their Support Confidant.
  The intervention consists of (1) selection and invitation of a Support Confidant, (2) a face-to-face intervention between the Intervention Case Manager and the Index and Support Confidant, and (3) quarterly interactive mini-booster sessions delivered to the Index and Support Confidant via text or telephone, based on participant preference.
  At 12 months, Index participants in the experimental condition will be re-randomized to either continue receiving quarterly interactive mini-booster sessions or to stop receiving mini-boosters and return to treatment as usual.
  Interventions: Behavioral: Social Network Support Intervention
- Treatment as Usual Condition (No Intervention): Treatment as Usual is comprehensive and follows Department of Health and Human Services guidelines and local protocols on the provision of HIV primary care, which include scheduling one HIV primary care visit and lab tests (including viral load) once every six months, i.e., two HIV primary care visits per year. In addition, all sites provide standard case management and mental health and psychosocial support services to all patients.

INTERVENTIONS:
Behavioral: Social Network Support Intervention — The Social Network Support Intervention is an evidence-based, flexible, and tailored intervention that leverages existing social network members to promote retention in care and viral suppression among people living with HIV. The intervention consists of (1) selection and invitation of a Support Confidant, (2) a face-to-face intervention between the Intervention Case Manager and the Index and Support Confidant, and (3) quarterly interactive mini-booster sessions delivered to the Index and Support Confidant via text or telephone, based on participant preference.
  Arms: Social Network Support Intervention Condition

SUMMARY:
The goal of this Hybrid Type I effectiveness-implementation trial is to test an evidence-based, flexible, and tailored intervention that leverages existing social network members to promote retention in care and viral suppression among people living with HIV aged 18-49.

DETAILED DESCRIPTION:
This study is a Hybrid Type I effectiveness-implementation trial of an evidence-based, flexible, and tailored intervention that leverages existing social network members to promote retention in care and viral suppression. The study will be conducted in Chicago, Illinois and Alabama, two high burden priority areas in the National Ending the HIV Epidemic Plan. Both retention in care and viral suppression are critical targets in ongoing efforts to eliminate HIV, as persons adherent to antiretrovirals are unlikely to transmit HIV, and retention in care allows for ongoing monitoring of viral load and the delivery of other important services, e.g., case management, mental health, and substance use treatment.

Most clinic-based strategies to improve Continuum of Care outcomes focus on newly created network members, e.g., support groups, peer navigators, or case managers. In contrast, we identify and activate organic Support Confidants (SC)-those people who can offer the types of social support that can help to navigate life's complexities, including the stressors of living with HIV. The intervention uses sociograms, highly engaging social network diagrams, to identify an ideally positioned Support Confidant. Once a Support Confidant is identified, the Index and their Support Confidant attend a single session, in-person intervention with a trained interventionist. The intervention uses the Information Motivation Behavioral Skills Model, Motivational Interviewing, and Cognitive Behavioral Theory to promote Continuum of Care-specific support in the Index-Support Confidant relationship.

This study will conduct a Hybrid Type I randomized controlled trial with N=600 participants living with HIV, who will be randomized to receive the intervention (n=300) or treatment as usual (n=300). In addition, 300 Support Confidants also will be enrolled. At 12-months post-intervention, we will re-randomize dyads to continue receiving mini-boosters (n=150) or return to treatment as usual (n=150). Data collection at baseline, 12, and 18 months will include surveys and electronic medical record (EMR) data. The study will be implemented in community-based clinics and academic-affiliated health centers in Chicago and in Birmingham and Huntsville, Alabama. To study implementation in each setting and geographic context, we will use the Consolidated Framework for Implementation Research as the determinant framework and Reach, Effectiveness, Adoption, Implementation, and Maintenance as the evaluation framework. The specific aims of the study are to:

Aim 1: Evaluate the (a) effectiveness of a social support intervention versus treatment as usual over 12 months with 600 people living with HIV ages 18-49 and (b) value of continuing to offer social support over another 6 months. The primary outcomes are retention in care and Viral Suppression, as measured by electronic medical record data on missed visit proportion and viral load.

Aim 2: Examine if intervention effects (a) vary between Chicago and Alabama, (b) are mediated by changes in the Index's level of motivational readiness, self-efficacy, and stigma expectancies, and (c) are moderated by mental health and substance use at the Index level.

Aim 3: Evaluate the implementation of the intervention using the Consolidated Framework for Implementation Research and the Reach, Evaluation, Adoption, Implementation and Maintenance frameworks. We will conduct surveys and focus groups with key stakeholders to assess the inner and outer settings, implementer and intervention characteristics, and multi-level process factors within the Consolidated Framework for Implementation Research. We will assess the following implementation outcomes for the study in each clinical setting and geographic context: Reach, Adoption, Implementation, and Maintenance.

If effective, the intervention has the potential to reduce HIV incidence by harnessing existing social support in the lives of people living with HIV, strengthening the public health impact of Treatment as Prevention. Thus, the research holds significant promise for addressing racial and geographic health disparities and will result in a sustainable, scalable program and implementation strategy that can be disseminated in HIV clinics nationwide.

ELIGIBILITY:
Inclusion Criteria for Index Participants:

* Aged 18-49 years old, inclusive
* Speak English
* Own a cell phone not shared with anyone else
* Have missed at least one HIV care scheduled visit or have not been virally suppressed in the past 24 months.
* Resides in Chicagoland, Illinois or Alabama

Exclusion Criteria for Index Men:

* If a participant fails to meet all inclusion criteria

Inclusion Criteria for Support Confidants:

* Index agrees to engage the Support Confidant
* Age 18 years or older
* Speaks English
* Owns a cell phone not shared with others
* Is not a romantic/sexual partner of the Index participant

Exclusion Criteria:

* Romantic/Sexual partners of Index participant
* Relationship strain or abuse present in Index-Support Confidant relationship

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Missed Visit Proportion | 18 months
  We count visits as scheduled (non-acute) visits to an antiretroviral prescribing provider. Missed Visit Proportion (MVP) is calculated as the proportion of total scheduled visits that are missed during the follow-up period. To permit longitudinal analyses, we shall also split the two-year follow-up period into eight three-month quarters and record, for each participant, whether he completed or missed his scheduled appointment during that quarter. Appointment and visit history to calculate MVP will be collected from each clinic's electronic medical record data.
Viral Suppression | 18 months
  Viral load (suppressed or not) will be measured in RNA copies/mL, with ≤200 copies/mL defined as viral suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Alida Bouris, PhD, Principal Investigator — University of Chicago; David S Batey, PhD, Principal Investigator — Tulane University
Locations (7):
- United States (7):
  - University of Alabama at Birmingham 1917 Clinic, Birmingham, Alabama
  - Birmingham AIDS Outreach, Birmingham, Alabama
  - Thrive Alabama, Huntsville, Alabama
  - Howard Brown Health, Chicago, Illinois
  - Chicago Center for HIV Elimination, Chicago, Illinois
  - Crown Family School of Social Work, Policy, and Practice at the University of Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be available to researchers outside of the study team.

REFERENCES:
- [Background] Bouris A, Jaffe K, Eavou R, Liao C, Kuhns L, Voisin D, Schneider JA. Project nGage: Results of a Randomized Controlled Trial of a Dyadic Network Support Intervention to Retain Young Black Men Who Have Sex With Men in HIV Care. AIDS Behav. 2017 Dec;21(12):3618-3629. doi: 10.1007/s10461-017-1954-8. PMID 29079949
- [Background] Bouris A, Voisin D, Pilloton M, Flatt N, Eavou R, Hampton K, Kuhns LM, Eder M, Schneider JA. Project nGage: Network Supported HIV Care Engagement for Younger Black Men Who Have Sex with Men and Transgender Persons. J AIDS Clin Res. 2013 Aug 31;4:10.4172/2155-6113.1000236. doi: 10.4172/2155-6113.1000236. PMID 24404408
- [Background] Cabral HJ, Tobias C, Rajabiun S, Sohler N, Cunningham C, Wong M, Cunningham W. Outreach program contacts: do they increase the likelihood of engagement and retention in HIV primary care for hard-to-reach patients? AIDS Patient Care STDS. 2007;21 Suppl 1:S59-67. doi: 10.1089/apc.2007.9986. PMID 17563291
- [Background] Centers for Disease Control and Prevention. Estimated HIV incidence and prevalence in the United States, 2010-2015. HIV Surveillance Supplemental Report 2018;23(No. 1). http://www.cdc.gov/hiv/library/reports/hiv-surveillance.html. Published March 2018. Accessed [1 Dec 2022].
- [Background] Craw JA, Gardner LI, Marks G, Rapp RC, Bosshart J, Duffus WA, Rossman A, Coughlin SL, Gruber D, Safford LA, Overton J, Schmitt K. Brief strengths-based case management promotes entry into HIV medical care: results of the antiretroviral treatment access study-II. J Acquir Immune Defic Syndr. 2008 Apr 15;47(5):597-606. doi: 10.1097/QAI.0b013e3181684c51. PMID 18285714
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Department of Health and Human Services. Ending the HIV Epidemic: A Plan for America. 2019; https://www.hhs.gov/sites/default/files/ending-the-hiv-epidemic-fact-sheet.pdf.
- [Background] Diggle P, Liang K, Zeger S. Analysis of Longitudinal Data: Oxford Statistical Science Series. 1994.
- [Background] Eisinger RW, Dieffenbach CW, Fauci AS. HIV Viral Load and Transmissibility of HIV Infection: Undetectable Equals Untransmittable. JAMA. 2019 Feb 5;321(5):451-452. doi: 10.1001/jama.2018.21167. No abstract available. PMID 30629090
- [Background] Fauci AS, Redfield RR, Sigounas G, Weahkee MD, Giroir BP. Ending the HIV Epidemic: A Plan for the United States. JAMA. 2019 Mar 5;321(9):844-845. doi: 10.1001/jama.2019.1343. No abstract available. PMID 30730529
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Fitzmaurice GM, Laird NM, Ware JH. Applied longitudinal analysis. Vol 998: John Wiley & Sons; 2012.
- [Background] Garamszegi LZ. Comparing effect sizes across variables: generalization without the need for Bonferroni correction. Behavioral Ecology. 2006;17(4):682-687.
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Higa DH, Marks G, Crepaz N, Liau A, Lyles CM. Interventions to improve retention in HIV primary care: a systematic review of U.S. studies. Curr HIV/AIDS Rep. 2012 Dec;9(4):313-25. doi: 10.1007/s11904-012-0136-6. PMID 22996171
- [Background] Hogan B, Carrasco JA, Wellman B. Visualizing Personal Networks: Working with Participant-aided Sociograms. Field Methods. 2007;19(2):116-144.
- [Background] Hoots BE, Finlayson TJ, Wejnert C, Paz-Bailey G; National HIV Behavioral Surveillance (NHBS) Study Group. Updated Data on Linkage to Human Immunodeficiency Virus Care and Antiretroviral Treatment Among Men Who Have Sex With Men-20 Cities, United States. J Infect Dis. 2017 Oct 17;216(7):808-812. doi: 10.1093/infdis/jix007. PMID 28368493
- [Background] Jiang H, Kulkarni PM, Mallinckrodt CH, Shurzinske L, Molenberghs G, Lipkovich I. Covariate Adjustment for Logistic Regression Analysis of Binary Clinical Trial Data. Statistics in Biopharmaceutical Research. 2017;9(1):126-134.
- [Background] Liang K-Y, Zeger SL. Longitudinal data analysis using generalized linear models. Biometrika. 1986;73(1):13-22.
- [Background] McCullagh P, Nelder J. Generalized linear models., 2nd edn.(Chapman and Hall: London). Standard book on generalized linear models. 1989.
- [Background] Naar-King S, Templin T, Wright K, Frey M, Parsons JT, Lam P. Psychosocial factors and medication adherence in HIV-positive youth. AIDS Patient Care STDS. 2006 Jan;20(1):44-7. doi: 10.1089/apc.2006.20.44. PMID 16426155
- [Background] Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents with HIV. Department of Health and Human Services. Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV. Available at http://www.aidsinfo.nih.gov/ContentFiles/ AdultandAdolescentGL.pdf.
- [Background] Starace F, Massa A, Amico KR, Fisher JD. Adherence to antiretroviral therapy: an empirical test of the information-motivation-behavioral skills model. Health Psychol. 2006 Mar;25(2):153-62. doi: 10.1037/0278-6133.25.2.153. PMID 16569106
- [Background] Valeri L, Vanderweele TJ. Mediation analysis allowing for exposure-mediator interactions and causal interpretation: theoretical assumptions and implementation with SAS and SPSS macros. Psychol Methods. 2013 Jun;18(2):137-50. doi: 10.1037/a0031034. Epub 2013 Feb 4. PMID 23379553
- [Background] VanderWeele TJ, Vansteelandt S. Mediation Analysis with Multiple Mediators. Epidemiol Methods. 2014 Jan;2(1):95-115. doi: 10.1515/em-2012-0010. PMID 25580377
- [Background] VanderWeele TJ, Tchetgen Tchetgen EJ. Mediation analysis with time varying exposures and mediators. J R Stat Soc Series B Stat Methodol. 2017 Jun;79(3):917-938. doi: 10.1111/rssb.12194. Epub 2016 Jun 27. PMID 28824285
- [Background] Vittinghoff E, Sen S, McCulloch CE. Sample size calculations for evaluating mediation. Stat Med. 2009 Feb 15;28(4):541-57. doi: 10.1002/sim.3491. PMID 19065627
- [Background] White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Stat Med. 2011 Feb 20;30(4):377-99. doi: 10.1002/sim.4067. Epub 2010 Nov 30. PMID 21225900

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT05723653/SAP_000.pdf